CLINICAL TRIAL: NCT06676332
Title: Effect of Multisensory Motor Imagery Training on Muscle Performance and Coordination in Children With Spastic Diplegia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mayada Ibraheem Elmahdy, Effect of multisensory motor imagery training on muscle performance and coordination in children with spastic diplegia, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 005278
Record Dates: First submitted 2024-09-09; First posted 2024-11-06 (Actual); Last update posted 2025-02-18 (Actual); Status verified 2025-02

CONDITIONS: Spastic Diplegia; Motor Imagery
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- control (Sham Comparator): traditional physical therapy program
  Interventions: Other: traditional physical therapy
- motor imagery (Experimental): multisensory motor imagery training plus the traditional physical therapy program
  Interventions: Other: motor imagery training; Other: traditional physical therapy

INTERVENTIONS:
Other: motor imagery training — Children in the study group will receive multisensory motor imagery training program 45 minutes. The training protocol consists of several parts that will be run through every training session according to Kumar et al. (2016):
  * Watching videos of selected multisensory motor skills for 10 minutes.
  * Mental rehearsal of these motor skills 10 minutes.
  * Overt practice of the multisensory motor skills for 25 minutes. On the videos, the performance of the skill by a child aged 8-12 years will be shown. All the exercises will be looped to repeat for six to seven times. While projecting the video on the laptop screen, it will be ensured that the children are in a comfortable seating position and the screen is in their visual field. Repetition of the exercises was based on their ability which could be a minimum of five repetitions per session to a maximum of ten repetitions per exercise session.
  Other Names: mental rehearsal exercises
  Arms: motor imagery
Other: traditional physical therapy — traditional physical therapy training program

SUMMARY:
PURPOSE:

The current study aims to:

* Determine the effect of multisensory motor imagery training on muscle performance including (peak torque, work, power) of trunk and knee flexors and extensors in children with spastic diplegia.
* Determine the effect of multisensory motor imagery training on coordination, strength and agility in children with spastic diplegia.

BACKGROUND: Multisensory motor imagery training has an effect on muscle performance and coordination in children with spastic diplegia

HYPOTHESES: There will be no effect of multisensory motor imagery training on muscle performance, coordination and strength and agility in children with spastic diplegic CP.

RESEARCH QUESTION: Is there an effect of multisensory motor imagery training on coordination, strength and agility in children with spastic diplegia?

ELIGIBILITY:
Inclusion Criteria:

* Their age will be ranged from 8-12 years.
* Mild degree of spasticity ranged from 1 to 1+ according to Modified Ashworth Scale
* Their motor function will be at level I and II according to Gross Motor Function Classification System GMFCS
* They will be able to follow instructions during evaluation and treatment.

Exclusion Criteria:

* - Cardiovascular or respiratory disorders.
* Botulinium muscular injection in the last 6 months
* Surgical interference in lower limbs and/or spine.
* Muscloskeletal problems or fixed deformities in the spine and/or lower extremities.
* Seizures.
* Visual or hearing impairment

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2024-11-16 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-05 (Estimated)

PRIMARY OUTCOMES:
muscle performance | through study completion average 3 months
  muscle performance of knee and trunk muscles will be assessed by Isokinetic dynamometer
coordination | through study completion average 3 months
  coordination ill be assessed using BOT-2

CONTACTS AND LOCATIONS:
Locations (1):
- Mayada Elshahawy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided